CLINICAL TRIAL: NCT01841723
Title: A Multicenter Phase 2 Study of the Bruton's Tyrosine Kinase Inhibitor PCI-32765 (Ibrutinib) for Treatment of Relapsed Hairy Cell Leukemia
Brief Title: Ibrutinib in Treating Patients With Relapsed Hairy Cell Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00826; NCI-2013-00826 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012C0139; P131378; OSU-12200; 9268 (Other: Ohio State University Comprehensive Cancer Center); 9268 (Other: CTEP); N01CM00039 (NIH); P30CA016058 (NIH); U01CA076576 (NIH); UM1CA186712 (NIH); NCT01981512 (obsolete NCT alias)
Record Dates: First submitted 2013-04-24; First posted 2013-04-26 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Hairy Cell Leukemia; Hairy Cell Leukemia Variant; Recurrent Hairy Cell Leukemia; Recurrent Hairy Cell Leukemia Variant
MeSH Terms: conditions — Leukemia, Hairy Cell | interventions — Specimen Handling; Biopsy; ibrutinib; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (ibrutinib) (Experimental): Patients receive ibrutinib PO QD on days 1-28. Cycles repeat every 28 days for up to 8 cycles if lack of response to therapy, up to 12 cycles if failure to achieve an objective response (CR/PR), or continually at per physician discretion in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo bone marrow aspiration and biopsy, blood sample collection, and CT or ultrasound throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Ibrutinib; Procedure: Ultrasound Imaging

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration and biopsy
Procedure: Bone Marrow Biopsy — Undergo bone marrow aspiration and biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA 032765; CRA-032765; CRA032765; Imbruvica; PCI 32765; PCI-32765; PCI32765
Procedure: Ultrasound Imaging — Undergo ultrasound
  Other Names: 2-Dimensional Grayscale Ultrasound Imaging; 2-Dimensional Ultrasound Imaging; 2D-US; Ultrasonography; Ultrasound; Ultrasound Test; Ultrasound, Medical; US

SUMMARY:
This phase II trial studies how well ibrutinib works in treating patients with hairy cell leukemia that has returned after a period of improvement. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the overall response rate (complete response [CR] and partial response [PR]) of hairy cell leukemia (HCL) at 32 weeks after beginning therapy with single-agent ibrutinib.

SECONDARY OBJECTIVES:

I. To characterize the toxicity and tolerability of single-agent ibrutinib when administered to patients with HCL.

II. To characterize the progression-free (PFS) and overall survival (OS) of single-agent ibrutinib when administered to patients with HCL.

III. To determine the rate of molecular remission (minimal residual disease [MRD]-negative CR) among all patients, defined as resolution of all detectable disease below the limits of detection by immunohistochemistry and/or 4-color flow cytometry assay at 32 weeks after beginning ibrutinib therapy.

IV. To characterize immunologic outcomes during single agent ibrutinib administration.

V. To explore the effect of ibrutinib (PCI-32765) on traditional and new biomarkers in HCL including:

Va. Confirmation of expression BRAFV600E in leukemia cells Vb. Pharmacodynamic effects of BTK inhibition on phosphorylated (phospho) ERK regulation, as well as other potential protein kinase targets of ibrutinib (exploratory) Vc. Serum soluble IL-2 receptor correlation with response to ibrutinib therapy Vd. Documentation of and quantification of minimal residual disease following maximal response, with flow cytometric analysis and immunohistochemical stains of the bone marrow, as predictors of remission duration after ibrutinib therapy.

OUTLINE:

Patients receive ibrutinib orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days for up to 8 cycles if lack of response to therapy, up to 12 cycles if failure to achieve an objective response (CR/PR), or continually at per physician discretion in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo bone marrow aspiration and biopsy, blood sample collection, and computed tomography (CT) or ultrasound throughout the study.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of hairy cell leukemia or variant according to World Health Organization (WHO) criteria with any of the following indications for therapy:

  * Hemoglobin < 11 g/dL
  * Platelet count < 100,000/mL
  * Absolute neutrophil count < 1,000/mL
  * Progressive or symptomatic splenomegaly or hepatomegaly
  * Enlarging lymphadenopathy >= 2 cm
  * Absolute lymphocyte count > 5,000/mL
  * Disease related constitutional symptoms consisting of unexplained weight loss exceeding 10% of body weight over the preceding 6 months, Cancer Therapy Evaluation Program (CTEP) active version of the Common Terminology Criteria for Adverse Events (CTCAE) grade 2 or 3 fatigue, fevers > 100.5 degrees Fahrenheit (F) or night sweats for greater than 2 weeks without evidence of infection
* Patients with classic hairy cell leukemia may receive therapy under the following conditions:

  * After at least 1 prior purine nucleoside analog-containing regimen (fludarabine, pentostatin, or cladribine), or
  * Relapsed or de novo disease if deemed medically unfit for therapy with a purine nucleoside analog

    * Because there is no recognized standard of care for patients with variant hairy cell leukemia, both previously treated and previously untreated patients with this diagnosis will be eligible
* Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of ibrutinib in patients < 18 years of age, children are excluded from this study, but may be eligible for future pediatric trials
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 12 months
* Creatinine =< 2.0 mg/dL, and/or creatinine clearance (estimated glomerular filtration rate [GFR] [Cockcroft-Gault]) >= 30 mL/min
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (unless disease related or due to Gilbert's disease)
* Aspartate aminotransferase (AST) =< 3.0 x ULN (unless disease related)
* Prothrombin time (PT)/international normalized ratio (INR) < 1.5 x ULN
* Partial thromboplastin time (PTT) (activated partial thromboplastin time [aPTT]) < 1.5 x ULN
* Because patients with HCL are typically pancytopenic at presentation for treatment, patients will be eligible without respect to baseline peripheral blood cell counts if they otherwise meet inclusion criteria
* The effects of ibrutinib on the developing human fetus are unknown; for this reason, and because tyrosine kinase inhibitors may be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry; female patients who are of non-reproductive potential (i.e., post-menopausal by history - no menses for >= 1 year; or history of hysterectomy; or history of bilateral tubal ligation; or history of bilateral oophorectomy); female patients of childbearing potential must have a negative serum pregnancy test upon study entry; male and female patients who agree to use highly effective methods of birth control (e.g., condoms, implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], complete sexual abstinence, or sterilized partner) during the period of therapy and for 90 days after the last dose of study drug; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Chemotherapy =< 21 days prior to first administration of study treatment and/or monoclonal antibody =< 6 weeks prior to first administration of study treatment
* Patients who are receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition as ibrutinib
* Ibrutinib is extensively metabolized by CYP3A4/5; patients who received a strong cytochrome P450 (CYP) 3A inhibitor within 7 days prior to the first dose of ibrutinib or patients who require continuous treatment with a strong CYP3A inhibitor; therefore, any medications or substances that are strong inhibitors of CYP3A4/5 should be discontinued; patients unable to change these medications must be excluded from participation; because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list; medical reference texts such as the Physicians' Desk Reference may also provide this information; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements; recent infections requiring systemic treatment need to have completed therapy > 14 days before the first dose of study drug
* Pregnant women are excluded from this study because ibrutinib is a tyrosine kinase inhibitor with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ibrutinib, breastfeeding should be discontinued if the mother is treated with ibrutinib
* Human immunodeficiency virus (HIV)-positive patients will be eligible unless they have been previously diagnosed with an acquired immune deficiency syndrome (AIDS)-defining illness
* Patients who require anticoagulation with warfarin (Coumadin) or who have taken warfarin within 28 days prior to enrollment are not eligible due to a potential increased risk of hemorrhage; patients who are currently taking vitamin K antagonists are also ineligible for this study
* Patients requiring daily corticosteroids at a prednisone equivalent of >= 20 mg daily should not be enrolled; if corticosteroids can be discontinued (or reduced to < 20 mg per day of prednisone or equivalent), the discontinuation or dose reduction should be done at least 7 days prior to first dose
* Prior exposure to a Bruton's tyrosine kinase (BTK) inhibitor
* Major surgery within 4 weeks of first dose of study drug
* A history of prior malignancy, with the exception of the following:

  * Malignancy treated with curative intent and with no evidence of active disease present for more than 3 years prior to screening, and felt to be at low risk for recurrence by the treating physician
  * Adequately treated non-melanomatous skin cancer or lentigo maligna melanoma without current evidence of disease
  * Adequately treated cervical carcinoma in situ without current evidence of disease
* Currently active clinically significant cardiovascular disease such as: uncontrolled arrhythmia, congestive heart failure, or class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification or history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to first dose with study drug
* Patient is unable to swallow capsules, or has disease significantly affecting gastrointestinal function or resection of the stomach or small bowel, or symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment
* Serologic status reflecting active hepatitis B or C infection; patients that are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody must have a negative polymerase chain reaction (PCR) prior to enrollment; (PCR positive patients will be excluded)
* Concurrent systemic immunosuppressant therapy other than corticosteroids (e.g., cyclosporine A, tacrolimus, etc.) within 28 days of the first dose of study drug
* Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug
* Unresolved toxicities from prior anti-cancer therapy, defined as having not resolved to Common Terminology Criteria for Adverse Event (CTCAE, version 5), grade =< 1, or to the levels dictated in the inclusion/exclusion criteria with the exception of alopecia
* Known bleeding disorders (e.g., von Willebrand's disease) or hemophilia
* Unwilling or unable to participate in all required study evaluations and procedures
* Currently active, clinically significant hepatic impairment (>= moderate hepatic impairment according to the National Cancer Institute [NCI]/Child Pugh classification)
* Incarceration at time of enrollment; prisoners will be excluded from enrollment; subjects who become incarcerated after starting study treatment will be allowed to continue in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2013-04-30 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (complete response [CR] and partial response [PR]) | 32 weeks
  Calculated as the proportion of patients who achieve a PR or CR to therapy within the first 32 weeks of therapy divided by the total number of evaluable patients.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 30 days after treatment
  Frequency and severity of adverse events and tolerability of the regimen in each of the patient groups will be collected and summarized by descriptive statistics and will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Progression-free survival | From the date of study registration to the date of event or the date of last follow-up if no event has occurred, assessed up to 3 years
  Kaplan-Meier curves will be used to estimate overall survival and time to next treatment.
Overall survival | From the date of study registration to the date of event or the date of last follow-up if no event has occurred, assessed up to 3 years
  Kaplan-Meier curves will be used to estimate overall survival and time to next treatment.
Rate of molecular remission (minimal residual disease [MRD]-negative CR) | Up to 32 weeks
  Defined as resolution of all detectable disease below the limits of detection by immunohistochemistry and 4-color flow cytometry assay will be examined.
Immunologic outcomes during single agent ibrutinib administration | Up to 12 months
Expression BRAFV600E in hairy cell leukemia cells | Baseline
  Markers will be summarized univariately in a quantitative manner and also summarized by clinical outcome group (e.g. responders vs. not). Graphical analyses will be largely used to assess potential patterns and relationships; e.g. side-by-side boxplots to assess differences in continuous marker levels between those with vs. without the clinical improvement.
Protein kinase regulation | Up to day 29 (day 1 of cycle 2)
  Pharmacodynamic effects of BTK inhibition on phosphorylated ERK regulation, as well as other possible protein kinase targets of ibrutinib including B lymphoid tyrosine kinase and BMX non-receptor tyrosine kinase/Etk will be assessed.
Serum soluble IL-2 receptor level | Up to 3 years
  Markers will be summarized univariately in a quantitative manner and also summarized by clinical outcome group (e.g. responders vs. not). Graphical analyses will be largely used to assess potential patterns and relationships; e.g. side-by-side boxplots to assess differences in continuous marker levels between those with vs. without the clinical improvement.
MRD level following maximal response | Up to 30 days after completing study treatment
  Will be with flow cytometric analysis and immunohistochemical stains of the bone as predictor of remission duration after ibrutinib therapy.

OTHER OUTCOMES:
Pharmacokinetic (PK) parameters | Predose, 0.5, 1, 2, 4, 6, and 24 hours post-dose on days 1 and 8 of cycle 1 and predose and 2 hours on days 15 and 22 of cycle 1 and day 1 of cycle 2
  Computed using non-compartmental and compartmental methods. Graphical analyses will be used as well as repeated measure models (linear or nonlinear mixed models, generalized estimating equation) to assess the PK markers in relation to clinical treatment outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Kerry A Rogers, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (5):
- United States (5):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - M D Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Rogers KA, Andritsos LA, Wei L, McLaughlin EM, Ruppert AS, Anghelina M, Blachly JS, Call T, Chihara D, Dauki A, Guo L, Ivy SP, James LR, Jones D, Kreitman RJ, Lozanski G, Lucas DM, Ngankeu A, Phelps M, Ravandi F, Schiffer CA, Carson WE, Jones JA, Grever MR. Phase 2 study of ibrutinib in classic and variant hairy cell leukemia. Blood. 2021 Jun 24;137(25):3473-3483. doi: 10.1182/blood.2020009688. PMID 33754642